CLINICAL TRIAL: NCT06212193
Title: Early Feasibility Study (EFS) to Assess the Safety and Performance of the Innoventric Trillium™ Stent Graft in the Treatment of Severe or Greater Tricuspid Regurgitation (TR)
Brief Title: Innoventric Trillium™ Stent Graft Early Feasibility Study (EFS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Innoventric LTD (Industry)
Collaborators: Innoventric Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLD-048
Record Dates: First submitted 2023-12-20; First posted 2024-01-18 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-11

CONDITIONS: Tricuspid Regurgitation; Tricuspid Regurgitation Functional
Keywords: Tricuspid valve; Transcatheter; Tricuspid Regurgitation; Tricuspid valve insufficiency
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Innoventric Trillium™ Stent Graft (Experimental): Transcatheter cross-caval tricuspid valve replacement with the Innoventric Trillium™ Stent Graft
  Interventions: Device: Trillium™

INTERVENTIONS:
Device: Trillium™ — Trillium™ Stent Graft for Cross-Caval Tricuspid Valve Replacement

SUMMARY:
Early Feasibility Study to evaluate the safety and performance of the Innoventric Trillium™ Stent Graft in the treatment of severe or greater tricuspid regurgitation (TR).

DETAILED DESCRIPTION:
Prospective, single arm, multi-center, Early Feasibility Study (EFS) to assess the safety and performance of the Innoventric Trillium™ Stent Graft in the treatment of severe or greater tricuspid regurgitation (TR).

Up to fifteen (15) patients at up to 10 US investigational sites and 3 German investigational sites will be enrolled. All enrolled study patients will be assessed at baseline, during the procedure, at discharge, and after 1 month, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years following the index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient has clinically significant TR graded as severe or greater
* Peak central venous pressure of ≥ 15mmHg
* Patient has NYHA functional classification of III or IV
* Patient is not eligible for standard-of-care surgical or interventional therapy or has refused standard-of-care surgical and interventional therapy or has received standard-of-care TR therapy and remains symptomatic

Exclusion Criteria:

Patients will be excluded from participation if ANY of the following criteria apply:

* Severe RV dysfunction defined by TAPSE, RVEF, or RVFAC.
* Anatomical suitability according to CT scan.
* Systolic Pulmonary Artery Pressure > 65mmHg
* Moderate or more mitral valve stenosis
* Greater than moderate mitral valve regurgitation or aortic valve stenosis/regurgitation
* Moderate mitral valve regurgitation combined with moderate aortic valve stenosis/regurgitation
* Kidney dysfunction with estimated Glomerular Filtration Rate (eGFR) < 35 ml/min/1.73 m2 within 60 days prior to the index procedure or patient is on chronic dialysis
* Liver cirrhosis or moderate or severe liver disease (Child-Turcotte-Pugh class B or C, or a score of 7 or higher)
* Thrombocytopenia (Platelet count< 80,000/mm3) or thrombocytosis (Platelet count > 750,000/mm3) within 14 days of the index procedure
* In the opinion of the Investigator or the study eligibility committee, the patient's life expectancy < 12 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Events [Safety endpoint] | at the end of the procedure, at discharge - typically within a week, and 30 days
  Rate of device or procedure-related Major Adverse Events (MAEs)
  And
  Rate of unplanned surgery or re-intervention due to a life-threatening device or procedure failure
Technical Performance | at the end of the procedure, at discharge - typically within a week, and 30 days
  Successful access, delivery, and retrieval of the Trillium™ delivery system, device is anchored both in SVC and IVC [at the end of the procedure]
  And
  No need for re-intervention due to device valve regurgitation or para-stent leak [at discharge, and 30 days]

SECONDARY OUTCOMES:
Rate of Major Adverse Events [Safety endpoint] | at 3 months, 6 months, 1, 2, 3, 4, and 5 years
  * Composite of all device or procedure-related MAEs [at 3 months, 6 months, 1, 2, 3, 4, and 5 years].
  * Device thrombosis, evaluated by Echocardiography [at 30 days, 6 months, 1, 2, and 4 years].
  * Device Migration as evaluated by Echocardiography or CMR [at 6 months]
Efficacy endpoint | at 30 days, 3-month, 6-month, 1-year, 2-year, 3-year, 4-year, and 5-year
  One or more of the following-
  * TR grade as measured on the device valves by Echocardiography, or reduction in peak CVP as measured by right heart catheterization [at the end of the procedure]
  * TR grade as measured on the device valves by Echocardiography [at 30 days, 6-month, 1-year, 2-year, and 4-year]
  * Rate of hospitalizations for HF [at 6-month, and 1-year]
  * HF functional class (NYHA) [at 30 days, 3-month, 6-month,1-year, 2-year, 3-year, 4-year, and 5-year]
  * Six-minute walk test (6MWT) [at 30 days, 6-month, 1-year, 2-year, and 4-year]
  * The Kansas City Cardiomyopathy Questionnaire (KCCQ) [at 30 days, 3-month, 6-month, 1-year, 2-year, 3-year, 4-year, and 5-year]
  * Patient Global Assessment (PGA) for Tricuspid Regurgitation Valve Treatment [at 30 days, 3-month, 6-month, 1-year, 2-year, 3-year, 4-year, and 5-year]

OTHER OUTCOMES:
Observational endpoint | at 30 days, 3 months, 6 months, 1, 2, 3, 4, and 5 years
  All-cause mortality

CONTACTS AND LOCATIONS:
Locations (12):
- United States (9):
  - Cardiovascular Institute of Los Robles Health System, Thousand Oaks, California
  - Ascension St. John, Detroit, Michigan
  - Mayo Clinic Hospital (Rochester), Rochester, Minnesota
  - Weill Cornell Medicine, New York, New York
  - Stony Brook Heart Institute, Stony Brook, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Lankenau Heart Institute, Philadelphia, Pennsylvania
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - University of Washington Medical Center, Seattle, Washington
- Germany (3):
  - University Medicine Mainz, Mainz, Rhineland-Palatinate
  - Helios Health Institute GmbH, Leipzig, Leipzig, Saxony
  - German Heart Center at Charité (DHZC), Berlin, State of Berlin